CLINICAL TRIAL: NCT04260282
Title: Exacerbations in Neutrophilic Asthma: Influence of Bronchial Microbiome
Brief Title: Microbiome and Exacerbations in Neutrophilic Asthma
Acronym: AsmaEx
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ANE-2020-04
Record Dates: First submitted 2020-01-23; First posted 2020-02-07 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Asthma; Microbiome; Exacerbation
MeSH Terms: conditions — Asthma | interventions — Bacterial Load

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Induced sputum Nasal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neutrophilic asthma: Patients with asthma diagnosed according to guidelines, with eosinophils <300/mm3 in blood and <3% in induced sputum
  Interventions: Diagnostic Test: Polymerase Chain Reaction (PCR) for viruses and bacteria in nasal swab; Diagnostic Test: Induced sputum microbiome
- Eosinophilic asthma: Patients with asthma diagnosed according to guidelines, with eosinophils >300/mm3 in blood and/or >3% in induced sputum
  Interventions: Diagnostic Test: Polymerase Chain Reaction (PCR) for viruses and bacteria in nasal swab; Diagnostic Test: Induced sputum microbiome

INTERVENTIONS:
Diagnostic Test: Polymerase Chain Reaction (PCR) for viruses and bacteria in nasal swab — PCR for viruses and bacteria in nasal swab
Diagnostic Test: Induced sputum microbiome — Microbiome in induced sputum

SUMMARY:
Neutrophilic asthma (NA) is the least known severe asthma phenotype. It is associated with more exacerbations, worse control and impaired lung function. One of its possible etiologies is bronchial infections. The study of bronchial microbiology and its relationship with exacerbations is a new line of research.

Objectives: 1) To analyze bronchial microbiome in patients with AN and non-neutrophilic (ANN), with frequent exacerbations and without exacerbations. 2) To relate the presence of bronchial infections with differences in the microbiome. 3) Correlate the characteristics of the microbiome with other evidence used in exacerbations.

Methods: Prospective study involving 40 non-smoking asthmatics without bronchiectasis (20 with AN and 20 with ANN). Of these, 10 in each group will have frequent exacerbations (>2 rounds of systemic steroids in the last year, of >3 days each) and 10 non- frequent exacerbations. AN will be defined as >65% neutrophils in stable phase sputum. All patients will have two stable visits in which clinical variables, asthma control, lung function and induced sputum samples will be collected (for analysis of bronchial inflammatory cell count and for the study of the microbiome by 16 subunit rRNA). Specific Immunoglobulin A (IgA) for Chlamydia Pneumoniae will be determined. In exacerbations, sputum samples will be collected for culture and nasopharyngeal smears for the study of major respiratory viruses and bacteria by multiple polymerase chain reaction.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 -80
* Confirmed diagnose of asthma
* Severe persistent asthma

Exclusion Criteria:

* Respiratory infection during the previous month
* Other significant lung disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe asthma according to guidelines, 18-80 years
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Differences between neutrophilic and non-neutrophilic asthma, with and without frequent exacerbations in bronchial microbiome using 16S rDNA sequencing | 6 months
  Qualitative and quantitative analysis of bronchial microbiome in patients including bacterial communities and major bacterial phyla in neutrophilic and non-neutrophilic asthma, with frequent exacerbations and without exacerbations.

SECONDARY OUTCOMES:
Changes in absolute and relative abundance using 16S rDNA sequencing of bronchial microbiota due to asthma exacerbations, in patients with neutrophilic and eosinophilic asthma | 1 year
  Influence of bronchial infections in qualitative and quantitative characteristics of lung microbiome. (Bacterial communities and major bacterial phyla)
Changes in absolute and relative abundance of bronchial microbiota over a year using 16S rDNA sequencing | 1 year
  Qualitative and quantitative changes of lung microbiome (Bacterial communities and major bacterial phyla)
Relationship between lung microbiome andlevels of specific immunoglobulin A of C. pneumoniae, PCR, and immunoglobulin G of aspergillus | 6 months
  Relationship between qualitative and quantitative characteristics of lung microbiome with levels of specific IgA C. pneumoniae, PCR, IgG aspergillus

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Crespo, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau. Carrer Mas Casanovas 90., Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddel HK, FitzGerald JM, Bateman ED, Bacharier LB, Becker A, Brusselle G, Buhl R, Cruz AA, Fleming L, Inoue H, Ko FW, Krishnan JA, Levy ML, Lin J, Pedersen SE, Sheikh A, Yorgancioglu A, Boulet LP. GINA 2019: a fundamental change in asthma management: Treatment of asthma with short-acting bronchodilators alone is no longer recommended for adults and adolescents. Eur Respir J. 2019 Jun 27;53(6):1901046. doi: 10.1183/13993003.01046-2019. Print 2019 Jun. No abstract available. PMID 31249014
- [Background] Plaza Moral V; Comite Ejecutivo de GEMA. [GEMA(4.0). Guidelines for Asthma Management]. Arch Bronconeumol. 2015 Jan;51 Suppl 1:2-54. doi: 10.1016/S0300-2896(15)32812-X. Epub 2015 Nov 30. No abstract available. Spanish. PMID 26707419
- [Background] Nair P, Aziz-Ur-Rehman A, Radford K. Therapeutic implications of 'neutrophilic asthma'. Curr Opin Pulm Med. 2015 Jan;21(1):33-8. doi: 10.1097/MCP.0000000000000120. PMID 25415406
- [Background] Wenzel SE, Szefler SJ, Leung DY, Sloan SI, Rex MD, Martin RJ. Bronchoscopic evaluation of severe asthma. Persistent inflammation associated with high dose glucocorticoids. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):737-43. doi: 10.1164/ajrccm.156.3.9610046. PMID 9309987
- [Background] Shaw DE, Berry MA, Hargadon B, McKenna S, Shelley MJ, Green RH, Brightling CE, Wardlaw AJ, Pavord ID. Association between neutrophilic airway inflammation and airflow limitation in adults with asthma. Chest. 2007 Dec;132(6):1871-5. doi: 10.1378/chest.07-1047. Epub 2007 Oct 9. PMID 17925424
- [Background] Brusselle GG, Vanderstichele C, Jordens P, Deman R, Slabbynck H, Ringoet V, Verleden G, Demedts IK, Verhamme K, Delporte A, Demeyere B, Claeys G, Boelens J, Padalko E, Verschakelen J, Van Maele G, Deschepper E, Joos GF. Azithromycin for prevention of exacerbations in severe asthma (AZISAST): a multicentre randomised double-blind placebo-controlled trial. Thorax. 2013 Apr;68(4):322-9. doi: 10.1136/thoraxjnl-2012-202698. Epub 2013 Jan 3. PMID 23291349
- [Background] Polosa R, Thomson NC. Smoking and asthma: dangerous liaisons. Eur Respir J. 2013 Mar;41(3):716-26. doi: 10.1183/09031936.00073312. Epub 2012 Aug 16. PMID 22903959
- [Background] Sutherland ER, Martin RJ. Asthma and atypical bacterial infection. Chest. 2007 Dec;132(6):1962-6. doi: 10.1378/chest.06-2415. PMID 18079229
- [Background] Uddin M, Nong G, Ward J, Seumois G, Prince LR, Wilson SJ, Cornelius V, Dent G, Djukanovic R. Prosurvival activity for airway neutrophils in severe asthma. Thorax. 2010 Aug;65(8):684-9. doi: 10.1136/thx.2009.120741. PMID 20685741
- [Background] Simpson JL, Baines KJ, Ryan N, Gibson PG. Neutrophilic asthma is characterised by increased rhinosinusitis with sleep disturbance and GERD. Asian Pac J Allergy Immunol. 2014 Mar;32(1):66-74. doi: 10.12932/AP0322.32.1.2014. PMID 24641293
- [Background] Green BJ, Wiriyachaiporn S, Grainge C, Rogers GB, Kehagia V, Lau L, Carroll MP, Bruce KD, Howarth PH. Potentially pathogenic airway bacteria and neutrophilic inflammation in treatment resistant severe asthma. PLoS One. 2014 Jun 23;9(6):e100645. doi: 10.1371/journal.pone.0100645. eCollection 2014. PMID 24955983
- [Background] Huang YJ, Nariya S, Harris JM, Lynch SV, Choy DF, Arron JR, Boushey H. The airway microbiome in patients with severe asthma: Associations with disease features and severity. J Allergy Clin Immunol. 2015 Oct;136(4):874-84. doi: 10.1016/j.jaci.2015.05.044. Epub 2015 Jul 26. PMID 26220531
- [Background] Blasi F. Atypical pathogens and respiratory tract infections. Eur Respir J. 2004 Jul;24(1):171-81. doi: 10.1183/09031936.04.00135703. PMID 15293621
- [Background] Frehn L, Jansen A, Bennek E, Mandic AD, Temizel I, Tischendorf S, Verdier J, Tacke F, Streetz K, Trautwein C, Sellge G. Distinct patterns of IgG and IgA against food and microbial antigens in serum and feces of patients with inflammatory bowel diseases. PLoS One. 2014 Sep 12;9(9):e106750. doi: 10.1371/journal.pone.0106750. eCollection 2014. PMID 25215528
- [Background] Rogers GB, Carroll MP, Serisier DJ, Hockey PM, Jones G, Bruce KD. characterization of bacterial community diversity in cystic fibrosis lung infections by use of 16s ribosomal DNA terminal restriction fragment length polymorphism profiling. J Clin Microbiol. 2004 Nov;42(11):5176-83. doi: 10.1128/JCM.42.11.5176-5183.2004. PMID 15528712